CLINICAL TRIAL: NCT03088319
Title: Chronic Stress Protection for Post-natal Depression Prevention: An Exploratory Study
Brief Title: Post-natal Depression and Chronic Stress
Acronym: serene
Status: Completed | Type: Observational
Sponsor: Institut de Recherche Biomedicale des Armees (Other Government)
Responsible Party: Principal Investigator, Marion Trousselard, senior researcher, Institut de Recherche Biomedicale des Armees
Other Study IDs: 2016-A00887-44
Record Dates: First submitted 2017-03-11; First posted 2017-03-23 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2018-08

CONDITIONS: Depression, Postpartum
Keywords: postnatal depression stress mindfulness allostatic load
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The risk of emergence of a post natal depression is based on an interaction between a maternal psychic vulnerability and a chronic environmental context of stress. The PND appears as a relevant model for studying the mechanisms of chronic stress and vulnerability to psychological pathologies.

This study aim to follow a cohort of pregnant women to determine the predictive psychobiological factors of the emergence of postnatal depression

DETAILED DESCRIPTION:
The prevalence of postnatal depression is high in civilian settings (20%). In mechanistic terms, the risk of emergence of a post natal depression is based on an interaction between a maternal psychic vulnerability and a chronic environmental context of stress. The post natal depression appears as a relevant model for studying the mechanisms of chronic stress and vulnerability to psychological pathologies.

* On the one hand, the repetition of stressors during pregnancy corresponds to a natural chronic stress model of several months and thus allows to study the biological cost of responses to repeated stresses, and the adaptive mechanisms leading to From functional drift to psychic dysfunction.
* On the other hand, isolated vulnerability factors characterize a mirroring psychological profile of a Mindfulness type of functioning. Mindfulness or full consciousness has been described as a state of consciousness which results from intentionally, at the present moment, without judging the experience that unfolds moment by moment. This psychological resource has been associated with resilient or even resilient psychic functioning.

This study aim to follow a cohort of pregnant women from the first trimester of pregnancies to 2 months after the delivery to determine the predictive psychobiological factors of the emergence of postnatal depression

ELIGIBILITY:
Inclusion Criteria:

* Physiological pregnancy
* Follow-up of pregnancy in a participating maternity
* Female over 18 years
* Affiliated to a social security scheme

Exclusion Criteria:

* Multiple pregnancy
* Psychiatric, neurological, or endocrine or autoimmune diseases
* Hormonal or psychotropic treatments

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: WOMEN DURING EARLY PREGNANCY
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
post natal depression | baseline at three 3 months of pregnancy and two months after labour delivery
  change in Edimbourg Post-Partum Depression scale at two months after labour delivery

SECONDARY OUTCOMES:
allostatic load as a composite index including blood GABA, BDNF and 8iso-Prostaglandins and capillary cortisol + heart rate variability index | baseline at three 3 months of pregnancy and two months after labour delivery
  change in allostatic load two months after labour delivery

OTHER OUTCOMES:
psychological functioning as a composite index including well-being, and stress control | baseline at three 3 months of pregnancy and two months after labour delivery
  change in psychological functioning two months after labour delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Marion Trousselard, Brétigny-sur-Orge, Not in US/Canada, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tharwat D, Trousselard M, Bales M, Sutter-Dallay AL, Fromage D, Spitz E, Dallay D, Harvey T, Welter E, Coatleven F, Cherier L, Teissedre F, Pouly JL, Dutheil F, Duffaud AM. Chronic Stress protection for postnatal dEpREssioN prEvention (SERENE): a protocol for an exploratory study. BMJ Open. 2018 May 3;8(5):e018317. doi: 10.1136/bmjopen-2017-018317. PMID 29724735